CLINICAL TRIAL: NCT06153381
Title: Herramienta de Procesamiento de Lenguaje Natural en Dispositivo móvil Inteligente Para Asegurar la Adherencia a la rehabilitación Domiciliaria en cirugías de Artroplastia Invertida de Hombro (NLP-PTAdherence)
Brief Title: Virtual Rehabilitation Assistant Via Instant Messaging Communication to Promote Adherence to Rehabilitation After Reverse Shoulder Replacement
Acronym: SIP_LaFe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Jose María Blasco Igual, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIP_LaFe
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot care (Experimental)
  Interventions: Other: Chatbot; Other: Standard car
- Standard care (Active Comparator)
  Interventions: Other: Standard car

INTERVENTIONS:
Other: Chatbot — Rehabilitation program based on standard care, but assisted via an instant messaging application using a personal smartphone
  Arms: Chatbot care
Other: Standard car — Rehabilitation program based on standard care, assisted with one education session plus informative brochure

SUMMARY:
reverse shoulder replacement surgery is performed to improve the functionality and reduce pain of the affected shoulder. Now, it is necessary to carry out an appropriate rehabilitation process to optimize surgical results. The lack of health resources makes it essential for the patient to work autonomously once hospital rehabilitation is completed. But lack of adherence is one of the main barriers to recovery

DETAILED DESCRIPTION:
The objective is to evaluate the effectiveness of a Chatbot that interacts with patients via instant messaging to supervise home rehabilitation and increase adherence. Conduct a feasibility study with a pilot sample

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing reverse shoulder replacement
* With a personal smartphone
* An instant messaging application installed
* Familiar with the use of such an application (i.e., at least three accessess per week)
* Able to write and read in the Spanish language

Exclusion Criteria:

* Condition, whether cognitive, neurological, integrative or musculoskeletal, that obviously prevents understanding or performing the exercises of the rehabilitation program or may pose a risk to the patient's health.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder disability | 0 weeks, 12 weeks
  This is measured with the Quick Dash questionnaire, a self-reported survey of 11 items designed to assess symptoms and ability to perform certain activities. At least 10 items should be answered to calculate a score. Each answer can be scored from one to five, and the average value is calculated, thus obtaining a score from one to five. Then, to express the score in percentages, 1 is subtracted from the result and then multiplied by 25. The higher the score, the greater the disability.

SECONDARY OUTCOMES:
Shoulder functionality | 0 weeks, 12 weeks
  measured with the Constant-Murley Score, a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively
Shoulder pain | 0 weeks, 12 weeks
  Assessed with a numeric pain rating scale, ranging from 0, the worst possible pain, to 10, no pain, with the question: What was your overall pain in the shoulder in the last week?
Quality of Life | 0 weeks, 12 weeks
  measured with the EQ-5D-5L quetionnaire, which essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Number of sessions of rehabilitation completed | 12 weeks
  Compliance with rehabilitation, measuring the number of sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain